CLINICAL TRIAL: NCT06896500
Title: Investigation Of The Effects Of Kegel Exercises On Vaginal Flatus Among Postpartum Women
Acronym: KEGEL-VF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: merve yilmaz menek (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor-Investigator, merve yilmaz menek, sponsor investigator, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-772.02-3326; E-10840098-772.02-3326 (Registry Identifier: Istanbul Medipol University Ethics Committee)
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pelvic Floor Awareness; Postpartum; Postpartum Pelvic Floor Function and Symptoms; Flatus
Keywords: kegel exercises; pelvic floor exercises; postpartum period; vaginal gas; vaginal flatus
MeSH Terms: conditions — Flatulence

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, randomized controlled trial with two arms: an experimental group performing Kegel exercises and a control group receiving no intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors were blinded to group allocation to prevent bias insubjective evaluations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegel Exercise Group (Experimental): Participants in this group performed Kegel exercises three times daily in different positions (supine, sitting, and standing) for three weeks, followed by a six-week home program. The exercises targeted both type I and type II muscle fibers with fast and slow contractions.
  Interventions: Behavioral: Kegel Exercises
- Control Group (No Intervention): Participants in this group did not perform any pelvic floor exercises and continued their routine postpartum activities. No intervention was applied

INTERVENTIONS:
Behavioral: Kegel Exercises — Kegel exercises performed three times daily in different positions (supine, sitting, and standing) for three weeks, followed by a six-week home program
  Arms: Kegel Exercise Group

SUMMARY:
Title: Investigation of the Effects of Kegel Exercises on Vaginal Flatus Among Postpartum Women

Brief Summary:

This study aims to evaluate the effectiveness of Kegel exercises in reducing vaginal flatus among postpartum women. Vaginal flatus, the involuntary passage of air through the vagina, is a common but often underreported pelvic floor dysfunction that can affect women's quality of life.

A total of 40 postpartum women were randomly assigned to an experimental group (performing Kegel exercises) or a control group (no intervention). The experimental group performed Kegel exercises three times daily in different positions for six weeks. Vaginal flatus frequency and bother scores were assessed using a validated questionnaire, and sexual quality of life was evaluated with the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12).

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to assess the effectiveness of Kegel exercises in reducing vaginal flatus among postpartum women. Vaginal flatus, the involuntary passage of air through the vagina, is a common but often overlooked pelvic floor dysfunction that can negatively impact women's quality of life.

A total of 40 postpartum women were recruited and randomly assigned to either the experimental group, which performed Kegel exercises, or the control group, which received no intervention. Participants in the experimental group were instructed to perform Kegel exercises three times daily in different positions (supine, sitting, and standing) over six weeks. The intervention focused on strengthening the pelvic floor muscles through a combination of fast and slow contractions targeting both Type I and Type II muscle fibers.

The primary outcome measures included vaginal flatus frequency and bother scores, which were assessed using a validated questionnaire before and after the intervention. Additionally, sexual quality of life was evaluated using the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12).

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 20-50,
* being postpartum at least 6 weeks after the last birth,
* having a complaint of vaginal flatus, and being willing to exercise

Exclusion Criteria:

* being over four months postpartum,
* current pregnancy,
* presence of pelvic infection,
* inability to indicate whether there is vaginal flatus,
* the presence of gynecological cancer.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only individuals who are biologically female and identify as femaleare eligible to participate
Enrollment: 40 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Vaginal Flatus Frequency Reduction | Baseline to at least 6 weeks postpartum
  The primary outcome is the change in vaginal flatus frequency, assessed via patient-reported questionnaire before and after the intervention. Smaller values indicate less flatus, while higher values signify an increase in flatus.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Kavasoglu Kaya, M.D., Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, I will not share IPD

REFERENCES:
- [Result] Lau HH, Su TH, Chen YY, Huang WC. The Prevalence of Vaginal Flatus in Women With Pelvic Floor Disorders and Its Impact on Sexual Function. J Sex Med. 2021 Mar;18(3):487-492. doi: 10.1016/j.jsxm.2020.12.008. Epub 2021 Jan 24. PMID 33504467
- [Result] Neels H, Pacquee S, Shek KL, Gillor M, Caudwell-Hall J, Dietz HP. Is vaginal flatus related to pelvic floor functional anatomy? Int Urogynecol J. 2020 Dec;31(12):2551-2555. doi: 10.1007/s00192-020-04371-9. Epub 2020 Jun 11. PMID 32529562
- Available data/document: Clinical Study Report: Ethics Committee Application — https://drive.google.com/file/d/19dj7wMiq4mPOobklxuHQObULyObAOvgc/view?usp=sharing
- Available data/document: Informed Consent Form: informed consent form — https://docs.google.com/document/d/1PuTtTRr_LxSuZvbzWyvw3EQZYQ0VyA7b/edit?usp=sharing&ouid=111712425749983896080&rtpof=true&sd=true
- Available data/document: Forms: Vaginal flatus status form — https://docs.google.com/document/d/1kFejPnvwa_N52yM8A2UKoAgZ3s1uPYuw/edit?usp=sharing&ouid=111712425749983896080&rtpof=true&sd=true
- Available data/document: Study Protocol: study main data — https://drive.google.com/file/d/1yPsrrEh2E2eVLPD-_QtWy8F0rgT0dM9g/view?usp=sharing